CLINICAL TRIAL: NCT05618873
Title: Comparative Effects of Flutter and Positive Expiratory Pressure on Chest Clearance and Dyspnea in Elderly Asthmatic Patients
Brief Title: Comparison of Flutter and PEP Mask on Chest Clearance, Dyspnea in Elderly Asthmatic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/ ALI HASSAN
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Asthma
Keywords: Flutter; PEP Mask; Chest Clearance; Dyspnea
MeSH Terms: conditions — Asthma; Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flutter device therapy (Experimental): The flutter was used as follows. Sitting with a straight back and the elbows supported on the table, the patient held the flutter horizontally. The patient inhaled deeply, held their breath for 2 or 3 s and then took the mouthpiece into the mouth and exhaled quietly yet quickly enough to activate the flutter. The patient had to keep their cheeks as stiff as possible. This procedure was repeated 15 times, following which the patient huffed three times and evacuated sputum by a voluntary cough. This sequence was repeated five times. The patient obtained the maximal vibration sensation by tilting the flutter upwards or downwards by a few degrees.
  Interventions: Device: Flutter device
- Positive Expiratory Pressure Mask (Experimental): The PEP-mask was used as follows. Sitting with a straight back and the elbows supported on the table, the patient pressed the mask against the face with both hands. After a quiet inhalation, a slow active exhalation followed. The exhalation was restricted by a resistance selected to cause a positive expiratory pressure of 8-12 cmH2O. The patient exhaled 15 times through the mask.
  Thereafter, the patient huffed three times and evacuated sputum by a voluntary cough. This sequence was repeated five times.
  Interventions: Device: positive expiratory pressure mask

INTERVENTIONS:
Device: Flutter device — The flutter was used as follows. Sitting with a straight back and the elbows supported on the table, the patient held the flutter horizontally. The patient inhaled deeply, held their breath for 2 or 3 s and then took the mouthpiece into the mouth and exhaled quietly yet quickly enough to activate the flutter. The patient had to keep their cheeks as stiff as possible. This procedure was repeated 15 times, following which the patient huffed three times and evacuated sputum by a voluntary cough. This sequence was repeated five times. The patient obtained the maximal vibration sensation by tilting the flutter upwards or downwards by a few degrees.
  Arms: flutter device therapy
Device: positive expiratory pressure mask — The PEP-mask was used as follows. Sitting with a straight back and the elbows supported on the table, the patient pressed the mask against the face with both hands. After a quiet inhalation, a slow active exhalation followed. The exhalation was restricted by a resistance selected to cause a positive expiratory pressure of 8-12 cmH2O. The patient exhaled 15 times through the mask.
  Thereafter, the patient huffed three times and evacuated sputum by a voluntary cough. This sequence was repeated five times.
  Arms: Positive Expiratory Pressure Mask

SUMMARY:
This study will be a Randomized controlled and will be conducted in Allied Hospital, Faisalabad. The study will be completed within the duration of 10 months. Convenience sampling study technique will be used to collect the data. The sample size of 30 patients will be taken in this study to find the effect of flutter and PEP mask therapy on chest clearance and dyspnea. Patients will be allocated randomly in two groups and 15 patients in each group. Group A will get flutter device therapy. Group B will get PEP mask treatment. A regular follow up visits to department and a final assessment was made at the end of last week by using questionnaire and resulting improvement was shown in results after completion. Data will be analyzed on SPSS25.

DETAILED DESCRIPTION:
This study will be a Randomized controlled and will be conducted in Allied Hospital, Faisalabad. The study will be completed within the duration of 10 months. Convenience sampling study technique will be used to collect the data. The sample size of 30 patients will be taken in this study to find the effect of flutter and PEP mask therapy on chest clearance and dyspnea. Patients will be allocated randomly in two groups and 15 patients in each group. Group A will get flutter device therapy. Group B will get PEP mask treatment. Treatment will be given to all the participants 3 sessionsin a week, or 2 weeks and post treatment evaluation will be done after every week. A regular follow up visits to department and a final assessment was made at the end of last week by using questionnaire and resulting improvement was shown in results after completion. Data will be analyzed on SPSS25.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis Of Asthma
* Both age above 40-60 years of age
* Both gender
* No previous surgery

Exclusion Criteria:

* Other pulmonary disease
* Neurological problems
* Rib fracture

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
ST. GEORGE'S RESPIRATORY QUESTINAIR | 2weeks
  The SGRQ is designed to measure health impairment in patients with asthma and COPD. Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Part I (Symptoms): several scales; Part II (Activity and Impacts): dichotomous (true/false) except last question (4-point Likert scale). Scores range from 0 to 100, with higher scores indicating more limitations.
PULMONARY FUNCTION TEST | 2weeeks
  Pulmonary function tests (PFTS) are an important tool in the investigation and monitoring of patients with respiratory pathology. The most basic test is spirometry. Spirometry is used to screen for diseases that affect lung volumes. It also is used to screen for diseases that affect the airways, such as COPD or asthma.
SPUTUM DIARY | 2weeks
  The diary card has a graded symptom score for dyspnea, sputum volume and sputum color. In addition, the card includes a score for patient well-being and documented all minor symptoms (cough, chest pain, cold, or flu-like symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Madiha younas, MS, Principal Investigator — riphah internationl university
Locations (1):
- Allied hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No